CLINICAL TRIAL: NCT06488677
Title: Influence of Social Determinants on Lifestyle Modification Adherence in People With Prediabetes: A Sequential Explanatory Mixed-Methods Study
Brief Title: Influence of Social Determinants on Lifestyle Modification Adherence in People With Prediabetes
Status: Not yet recruiting | Type: Observational
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/02723
Record Dates: First submitted 2024-06-12; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: PreDiabetes
Keywords: Healthy lifestyle; Social determinants of health; Prediabetes; Therapeutic adherence and compliance
MeSH Terms: conditions — Prediabetic State; Treatment Adherence and Compliance | interventions — Diet; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High adherence: Participants with high adherence to the lifestyle intervention
  Interventions: Behavioral: Lifestyle changes (diet and physical activity)
- Low adherence: Participants with low adherence to the lifestyle intervention
  Interventions: Behavioral: Lifestyle changes (diet and physical activity)

INTERVENTIONS:
Behavioral: Lifestyle changes (diet and physical activity) — Nurse-led telephone personalized dietary and PA advice

SUMMARY:
A sequential explanatory mixed-methods study analyzing the influence of social determinants on adherence to healthy lifestyle recommendations in individuals with prediabetes.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is a major risk factor for adult morbidity and mortality and represents a public health burden due to its rising global prevalence. T2D is preceded by prediabetes, a phase characterized by higher-than-normal blood glucose levels that do not reach the threshold required for a T2D diagnosis. It is estimated that 70% of people with prediabetes will eventually develop T2D, with a mean annual incidence rate ranging from 5% to 10%.

Importantly, socioeconomic status exacerbates the risk of developing chronic diseases such as T2D, as people from underprivileged social classes are significantly more susceptible to the development of the disease and its complications, when compared to the more privileged.

In fact, it has been observed that the risk of developing T2D extends beyond physiological factors. Social determinants (SD) such as age, gender, ethnicity, postal code, or socioeconomic status, and health beliefs are strong predictors of disease onset and progression. Populations with a low socioeconomic status (i.e., economically disadvantaged backgrounds, lower health literacy levels, lower educational status, and often, from ethnic and racial minorities), are known to experience reduced access to healthcare including health promotion programs. They also have lower adoption rates of health behaviors, such as physical activity (PA) and healthy diet, and thus be at increased risk of chronic diseases such as T2D, which finally increases their likelihood to suffer inequalities in mortality.

For all of the above, this study aims to explore the influence of SD on adherence behaviors in individuals with prediabetes included in the PREDIPHONE trial, using a mixed-methods sequential explanatory design. The findings from both the quantitative and qualitative phases will be integrated to offer a comprehensive understanding of the complex phenomenon of adherence.

ELIGIBILITY:
Inclusion Criteria:

* participants of the PREDIPHONE trial assigned to the intervention group and who complete the 9-month intervention period

Exclusion Criteria:

* Participants from the control group or those who withdrew from the trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with prediabetes included in the intervention arm of the PREDIPHOE randomized controlled trial.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to healthy lifestyle recommendations | at month 9 of the intervention period
  Adherence to healthy lifestyle recommendations measured through a composite index generated with data from 1) dietary adherence assessed using the 14-item PREDIMED Mediterranean Diet questionnaire and 2) physical activity adherence evaluated using the REGICOR Abbreviated Questionnaire.
Facilitators and barriers to adherence to lifestyle changes | at month 9 of the intervention period
  Facilitators and barriers to adherence to lifestyle changes such as social and family support, knowledge about one's health condition, health beliefs, and the patient-professional relationship

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carvalho-Azevedo A, Abbate M, Fresneda S, Arias-Fernandez M, Torres-Carballo M, Yanez AM, Moreno-Mulet C, Bennasar-Veny M. Influence of social determinants on lifestyle modification adherence in people with prediabetes: a sequential explanatory mixed-methods study protocol. Front Public Health. 2025 Jul 3;13:1591205. doi: 10.3389/fpubh.2025.1591205. eCollection 2025. PMID 40678653